CLINICAL TRIAL: NCT01524120
Title: Endoscopy and Endomicroscopy for Assessment of Mucosal Healing in Inflammatory Bowel Disease (IBD)
Status: Withdrawn | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: HN-0009
Record Dates: First submitted 2012-01-23; First posted 2012-02-01 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Mucosal healing
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies were taken from every patient for subsequent histological analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Crohn's disease (CD): Patients with CD and mucosal healing on endoscopy.
  Interventions: Device: Endoscopy (EPK-i, Pentax, Tokyo, Japan)
- Crohn's disease: Patients with CD and mucosal healing on endomicroscopy.
  Interventions: Device: Endomicroscopy (iCLE, Pentax, Tokyo, Japan)
- Ulcerative colitis (UC): Patients with UC and mucosal healing on endoscopy.
  Interventions: Device: Endoscopy (EPK-i, Pentax, Tokyo, Japan)
- Ulcerative colitis: Patients with UC and mucosal healing on endomicroscopy.
  Interventions: Device: Endomicroscopy (iCLE, Pentax, Tokyo, Japan)

INTERVENTIONS:
Device: Endoscopy (EPK-i, Pentax, Tokyo, Japan) — Patients will undergo white-light endoscopy. Any mucosal lesions will be recorded and findings will be compared to histopathological and clinical results.
  Groups: Crohn's disease (CD)
Device: Endomicroscopy (iCLE, Pentax, Tokyo, Japan) — Patients will undergo endomicroscopy. Data will be recorded and findings will be compared to histopathological and clinical results.
  Groups: Crohn's disease
Device: Endoscopy (EPK-i, Pentax, Tokyo, Japan) — Patients will undergo white-light endoscopy. Any mucosal lesions will be recorded and findings will be compared to histopathological and clinical results.
  Groups: Ulcerative colitis (UC)
Device: Endomicroscopy (iCLE, Pentax, Tokyo, Japan) — Patients will undergo endomicroscopy. Data will be recorded and findings will be compared to histopathological and clinical results.
  Groups: Ulcerative colitis

SUMMARY:
Inflammatory bowel disease (IBD) encompasses two major forms of chronic intestinal disorders, Crohn's disease and ulcerative colitis (UC). Diagnosis is based on several macroscopic and histologic features including patterns of inflammation, crypt abscesses and granulomas. Confocal laser endomicroscopy (CLE) is rapidly emerging as a valuable tool for gastrointestinal endoscopic imaging, enabling the endoscopist to obtain an "optical biopsy" of the gastrointestinal mucosa during the endoscopic procedure.

The main objective of this study is to determine endoscopic and endomicroscopic features of mucosal healing in patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-85 years
* Ability of subjects to understand character and individual consequences of clinical trial
* Subjects undergoing colonoscopy

Exclusion Criteria:

* Inability to provide written informed consent
* Severe Coagulopathy (Prothrombin time < 50% of control, Partial thromboplastin time > 50 s)
* Pregnancy or breast feeding
* Active gastrointestinal bleeding
* Residing in institutions (e.g. prison)
* Known allergy against fluorescein

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn´s disease and ulcerative colitis. Only patients with mucosal healing are included.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-04

PRIMARY OUTCOMES:
Mucosal healing | 3 years
  We will determine endoscopic (e.g. ulcera, erythema) and endomicroscopic features of mucosal inflammation (e.g. goblet cell depletion, leackage, microvessel density) in IBD in order to define new criteria of mucosal healing and to define factors of disease remission and relapse.

SECONDARY OUTCOMES:
Histologic correlation | 3 years
  Comparison of clinical and histopathological data with endoscopic and endomicroscopic findings to evaluate mucosal healing as a parameter of remission and relapse in patients with IBD.
Therapeutic effect | 3 years
  We will evaluate the effect of different therapeutic strategies (eg. anti-TNF treatment, corticosteroids) on characteristics of mucosal healing (e.g. goblet cell depletion, microvessels, leakage) and remission and relapse rate.

CONTACTS AND LOCATIONS:
Overall Officials: Markus F. Neurath, M.D., Ph.D., Principal Investigator — University of Erlangen-Nürnberg; Helmut Neumann, M.D., Ph.D., Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- University of Erlangen-Nuremberg, Erlangen, Germany